CLINICAL TRIAL: NCT05560165
Title: F-18 Sodium Fluoride PET/CT Guided Robotic Arm-assisted Pain Palliation in Chronic Nociceptive Low Backache
Brief Title: PET/CT Guided Robotic Arm-assisted Pain Palliation in Chronic Nociceptive Low Backache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Associate Professor, Department of Nuclear Medicine,, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2022/SPL-888
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2022-09

CONDITIONS: Chronic Low-back Pain; Nociceptive Pain
MeSH Terms: conditions — Nociceptive Pain | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/CT guided injection of combination of local anesthetic and steroids. (Experimental): The F-18 Sodium fluoride (NaF) dose will be administered intravenously and the F-18 NaF PET/CT images will be reviewed, and the target nociceptive site will be determined on the basis of increased focal tracer uptake. The joint accessibility, location, and relation with the nearby vital organs will be assessed. The injection will be assisted using a dedicated automated robotic arm system. A combination of corticosteroids and local anesthetic will be injected.
  Interventions: Procedure: F-18 sodium fluoride PET/CT guided robotic arm assisted injection of combination of local anesthetic and steroids

INTERVENTIONS:
Procedure: F-18 sodium fluoride PET/CT guided robotic arm assisted injection of combination of local anesthetic and steroids — A surgical aseptic approach will be followed for the procedure. Local anesthesia of the skin and soft tissue at the entry site will be achieved by 1% lignocaine. A 23G lumbar puncture needle will be introduced and the real-time final placement of the needle will be confirmed with low dose CT (40 mA) fused with pre-procedure PET images. After confirming the real-time position, the local anesthetic and steroid injection (0.5ml of 0.5% Bupivacaine per joint and a total dose of 80mg of Methylprednisolone acetate divided equally based on the number of joints to be injected) will be injected intraarticularly and periarticularly around the target joint through the lumbar puncture needle. The skin entry site will be compressed manually to achieve hemostasis. The same procedure will be repeated if multiple joints are to be injected. After the procedure, patient vitals will be observed for thirty minutes in the recovery area and discharged in stable condition.

SUMMARY:
A study to investigate the role of F-18 sodium fluoride in localizing the pain generator in participants with chronic nociceptive musculoskeletal low back ache and to study the use of PET/CT guided robotic arm assisted injection for targeted injection of a combination of corticosteroid and local anesthetic for pain palliation.

DETAILED DESCRIPTION:
Chronic pain in the lower back may be due to a variety of causes such as neuropathic causes, musculoskeletal causes, visceral causes, malignancy-related or primary pain where in there is no obvious cause of pain. Musculoskeletal pain usually affects the muscles, joints, bones or their surrounding soft tissue structures. These participants are usually evaluated with clinical examination and radiological imaging modalities such as computed tomography (CT) or Magnetic resonance imaging (MRI) to identify the pain generating site. The possible sites of involvement may include the sacroiliac joints, intervertebral facet joints, the vertebrae, the intervertebral discs, or the surrounding ligaments and muscles which may be apparent on imaging. They are usually started on oral analgesics such as Non-steroidal anti-inflammatory drugs as the first line of management. However, occasionally the patient may not respond to this line of management. In such cases, they may be treated with more potent analgesics or subjected to targeted local management of the pain-generating site with an injection of local anesthetics and corticosteroids. They are usually given at the site of tenderness following clinical examination or under image guidance using x-ray fluoroscopy or CT guidance. However, anatomical imaging modalities may not diagnose early stages of the disease or distinguish active from inactive disease. Bone scintigraphy with Tc-99m labeled phosphonates is known to diagnose and localize active sites of musculoskeletal pain. PET/CT with sodium fluoride is also useful in the same indication as it has similar pharmacodynamics to that of Tc-99m labeled phosphonates. The combination of image guidance with sodium fluoride PET/CT and the use of an automated robotic arm (ARA) can help in the targeted delivery of the local anesthetic and steroids to the nociceptive pain generating site. This study is intended to analyze the role of F-18 sodium fluoride in localizing the pain generator in participants with chronic nociceptive musculoskeletal low back ache and to study the use of PET/CT guided robotic arm assisted injection for targeted injection of steroid and local anesthetic for pain palliation in such participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic nociceptive low back ache (for more than three months) do not have adequate pain relief with oral analgesics.
* Participants who are ready to give written informed consent for the procedure

Exclusion Criteria:

* MRI showing the neuropathic cause of pain with spinal cord or nerve root compression.
* Extensive bone or joint destruction and displacement such as spondylolisthesis or compression fractures of the vertebra.
* Imaging, clinical and hematological findings suggestive of infective/ malignant pathology.
* Patients with deranged coagulation profile
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficacy of the procedure | Immediate - post procedure
  Diagnostic efficacy of F-18 sodium fluoride PET/CT for localizing the site of pain in patients with chronic nociceptive low back ache and assessing the reduction in pain following the procedure.The procedure will be believed as technically successful if there is a 50% decrease in the severity of pain following the procedure as assessed by the visual analogue score.
Treatment efficacy of the procedure | One month
  Treatment efficacy of injection of a combination of corticosteroid and local anesthetic intraarticularly following localization by F-18 sodium fluoride PET/CT in patients with chronic nociceptive low back ache. The visual analog score will be used to document the sustained reduction in pain for one month following the procedure.

SECONDARY OUTCOMES:
Safety of F-18 sodium fluoride PET/CT guided robotic arm assisted injection of local anesthetic and steroids. | Immediately following the procedure till 30 minutes and upto one month following the procedure
  To assess the immediate and delayed adverse effects following the procedure upto a period of one month.
Imaging based response assessment following F-18 sodium fluoride PET/CT guided robotic arm assisted injection of local anesthetic and steroids. | One month
  To quantify the resolution or decrease in the intensity of the tracer uptake in the target joints to assess the objective response to injection of local anesthetic and steroids by using F-18 sodium fluoride PET/CT at one month following injection. The images will be compared with those acquired at baseline to assess the response.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant information will be available from the principal investigator upon reasonable request for a period of five years from the date of completion of the study.
Supporting Information: Study Protocol, CSR
Time Frame: Five years from the date of completion of the study.
Access Criteria: Reasonable request to the principal investigator